CLINICAL TRIAL: NCT04008511
Title: Phase Ib/II Study of Regorafenib and XELOX Combination as 2nd Line Treatment in Metastatic Colorectal Cancer Patients
Brief Title: Regorafenib and XELOX as 2nd Line Treatment in Metastatic Colorectal Cancer
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: China Medical University, China (Other)
Collaborators: Liaoning Cancer Hospital & Institute (Other); The First People's Hospital of Jingzhou (Other)
Responsible Party: Principal Investigator, Yunpeng Liu, Director, China Medical University, China
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CLOG1901; IMPACT 20872 (Other Grant/Funding Number: Bayer Healthcare Company limited)
Record Dates: First submitted 2019-07-02; First posted 2019-07-05 (Actual); Last update posted 2019-07-05 (Actual); Status verified 2019-07

CONDITIONS: Metastatic Colorectal Cancer
Keywords: Metastatic Colorectal Cancer; Regorafenib; Second line; XELOX
MeSH Terms: conditions — Colorectal Neoplasms | interventions — regorafenib; Capecitabine; Oxaliplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Phase Ib: Regorafenib plus XELOX (Experimental): Phase Ib followed a Modified toxicity probability interval (mTPI) design to determine the maximum administered dose (MAD), there are 3 dose levels, and the dose level started from Group A:
  Group A: Regorafenib 120mg + XELOX; Group B: Regorafenib 160mg + XELOX; Group C: Regorafenib 80mg + XELOX. (Regorafenib qd po for 14 days, every 3 weeks; XELOX: Oxaliplatin 130 mg/m2 IV, day 1, Capecitabine 1000 mg/m2 bid po for 14 days)
  Interventions: Drug: Regorafenib; Drug: Capecitabine; Drug: Oxaliplatin
- Phase II: Regorafenib plus XELOX (Experimental): Regorafenib MAD qd po for 14 days, every 3 weeks, Oxaliplatin 130 mg/m2 IV on day 1, Capecitabine 1000 mg/m2 bid po for 14 days.
  Interventions: Drug: Regorafenib; Drug: Capecitabine; Drug: Oxaliplatin
- Phase II: XELOX (Active Comparator): Oxaliplatin 130 mg/m2 IV on day 1, Capecitabine 1000 mg/m2 bid po for 14 days.
  Interventions: Drug: Capecitabine; Drug: Oxaliplatin

INTERVENTIONS:
Drug: Regorafenib — Phase Ib Group A: Regorafenib 120mg + XELOX; Group B: Regorafenib 160mg + XELOX; Group C: Regorafenib 80mg + XELOX.
  Other Names: Stivarga
  Arms: Phase Ib: Regorafenib plus XELOX
Drug: Regorafenib — Phase II: Regorafenib MAD qd po for 14 days, every 3 weeks.
  Other Names: Stivarga
  Arms: Phase II: Regorafenib plus XELOX
Drug: Capecitabine — Capecitabine 1000 mg/m2 bid po for 14 days.
  Other Names: Xeloda
Drug: Oxaliplatin — Oxaliplatin 130mg/m2, day 1, every 3 weeks
  Other Names: ELOXATIN®

SUMMARY:
This is an interventional, randomized open-label, parallel-group, multicenter, dose escalation phase Ib/II study, to investigate the combination of Regorafenib and XELOX as 2nd line treatment in mCRC patients.

DETAILED DESCRIPTION:
This is a phase Ib/II trial, comprising Phase Ib and Phase II two parts. Phase Ib study is an open-label, single-arm, multicenter, dose escalation study of Regorafenib plus XELOX. In Phase Ib, max 15 patients(pts) could be enrolled based on the modified toxicity probability interval (mTPI) design. Phase II study is a randomized, open-label, parallel-group, multicenter study comparing Regorafenib + XELOX to XELOX alone. In phase II trial, a total of 39 patients will be recruited and randomized 2:1 into two groups, where 26 patients under Regorafenib + XELOX, and 13 patients under XELOX alone.

ELIGIBILITY:
Inclusion Criteria:

1. Sign a consent form
2. Age> 18 years <75 years
3. Pathological diagnosis as colorectal adenocarcinoma
4. Recurrence or metastatic disease
5. Metastatic colorectal cancer with disease progression after 1st line treatment by 5-Fu and Irinotecan
6. Measurable disease according to Response Evaluation Criteria in Solid Tumors (RECIST)
7. ECOG score 0-1 points
8. Life expectancy ≥3 months
9. Can provide more than 10 paraffin sections of tumor tissue
10. End of radiotherapy without or with non-targeted lesions> 4 weeks (only for use outside of the test site)
11. At least one measurable lesion (according to RECIST 1.1)
12. Previously treated radiotherapy lesions cannot be considered as target lesions, unless the radiotherapy lesions clear progress.
13. Alanine aminotransferase (ALT) and aspartate aminotransferase (AST)≤ 2.5 times the upper limit of normal (ULN), patients with liver metastases ≤ 5 times ULN
14. Serum albumin ≥ 3.0g / dL
15. Serum alkaline phosphatase (AKP) ≤2.5 times ULN
16. Total bilirubin <1.5mg / dL
17. Estimated creatinine clearance (CLcr) ≥ 30 mL/min as calculated using the Cockcroft-Gault equation
18. Lipase ≤ 1.5 x the ULN
19. Neutrophil absolute count (ANC) ≥ 1500 / mm3, hemoglobin (Hb)> 9g/dl, platelets> 100,000 / mm3
20. Pregnant or breast-feeding patients:

1) Women of childbearing potential and men must agree to use adequate contraception before entering the program until at least 8 weeks after the last study drug administration. The investigator or a designated associate is requested to advise the subject on how to achieve an adequate birth control. Adequate contraception is defined in the study as any medically recommended method (or combination of methods) as per standard of care.

2) Women of childbearing potential must have a blood or urine pregnancy test performed a maximum of 7 days before start of study treatment, and a negative result must be documented before start of study treatment

Exclusion Criteria:

1. Received oxaliplatin and capecitabine in the 1st line treatment
2. Cannot be orally administered
3. Subjects with brain metastases and / or cancerous meningitis.
4. Surgical treatment was performed within 4 weeks before enrollment (excluding diagnostic biopsies)
5. Non-healing wound, non-healing ulcer, or non-healing bone fracture
6. Patients with evidence or history of any bleeding diathesis, irrespective of severity
7. Any hemorrhage or bleeding event ≥ CTCAE Grade 3 within 4 weeks prior to the start of study medication.
8. Arterial or venous thrombotic or embolic events such as cerebrovascular accident (including transient ischemic attacks), deep vein thrombosis or pulmonary embolism within 6 months before the start of study medication (except for adequately treated catheter-related venous thrombosis occurring more than one month before the start of study medication)
9. Congestive heart failure ≥ New York Heart Association (NYHA) class 2
10. Uncontrolled cardiac arrhythmias
11. Ongoing infection > Grade 2 NCI CTCAE
12. Interstitial lung disease with ongoing signs and symptoms at the time of informed consent.
13. Known hypersensitivity to any of the study drugs, study drug classes, or excipients in the formulation.
14. Anti-tumor cytotoxic drug therapy, biologic medication (eg, monoclonal antibody), immunotherapy (eg, interleukin 2 or interferon), or other investigational drug therapy within 4 weeks prior to enrollment
15. Subjects with active tuberculosis (TB) who are on anti-TB treatment or who have received anti-TB treatment within 1 year prior to screening
16. Patients with complications requiring long-term use of immunosuppressive drug therapy or systemic or topical corticosteroids requiring immunosuppressive doses (prednisone or other equivalent hormones at doses> 10 mg / day)
17. Use of strong CYP3A4 inducers or inhibitors
18. In the first 4 weeks before the group vaccinated any anti-infective vaccine (such as influenza vaccine, varicella vaccine, etc.)
19. Pregnancy or lactation
20. 5 years with other malignancies, except for non-melanoma skin cancer
21. Persistent proteinuria > 3.5 g/24 hours measured by urine protein-creatinine ratio from a random urine sample (Grade 3, NCI-CTCAE v 5.0).
22. Human immunodeficiency virus (HIV) positive
23. Hepatitis B surface antigen (HBsAg) positive simultaneous detection of Hepatitis B virus (HBV) Deoxyribonucleic acid (DNA) copy number positive (quantitative detection ≥ 1000cps / ml)
24. Chronic hepatitis C blood screening positive [Hepatitis C virus (HCV) antibody positive]
25. No legal capacity
26. Any other disease or condition that the investigator considers may affect program adherence or affect the subject's signature of informed consent (ICF), or are not suitable for participating in this clinical trial.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Estimated)
Dates: Start 2019-07 (Estimated); Primary Completion 2023-03 (Estimated); Study Completion 2024-03 (Estimated)

PRIMARY OUTCOMES:
Maximum tolerated dose (MTD) | 6 weeks
  The MTD is defined as the highest dose that can be given so that toxicity probability is below the target toxicity PT=30%.
Progression-free survival (PFS) | 1 year
  PFS is defined as the time (days) from start of study treatment to date of first observed disease progression (investigator's radiological or clinical assessment) or death due to any cause, if death occurs before progression is documented.
Number of participants with treatment-related adverse events as assessed by CTCAE v5.0 | 3 years
  Safety and tolerability

SECONDARY OUTCOMES:
Disease control rate (DCR) | 3 years
  o DCR is defined as the percentage of patients, whose overall best response was not progressive disease.
Overall response rate (ORR) | 3 years
  o ORR is defined as the percentage of patients with complete response (CR) or partial response (PR).

CONTACTS AND LOCATIONS:
Overall Officials: Yunpeng Liu, M.D.,Ph.D., Principal Investigator — First Hospital of China Medical University
Locations (1):
- The First Hospital of China Medical University, Shenyang, Liaoning, China

IPD SHARING:
Plan to Share IPD: No